CLINICAL TRIAL: NCT01730339
Title: A Phase 2, Randomized, Double-blind, Within-subject, Placebo Controlled Study To Evaluate The Efficacy And Safety Of Pf 06473871 In Reducing Hypertrophic Skin Scarring
Brief Title: Safety and Efficacy Study of PF-06473871 to Reduce Hypertrophic Scars From Recurring Post-Revision Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: B5301001; 2012-004355-37 (EudraCT Number)
Record Dates: First submitted 2012-11-12; First posted 2012-11-21 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Reduction of Hypertrophic Skin Scarring
Keywords: Skin scarring; cicatrix; breast scar; hypertrophic scar
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Drug: PF-06473871
- Group 2 (Active Comparator)
  Interventions: Drug: PF-06473871

INTERVENTIONS:
Drug: PF-06473871 — Single dose administered by injection four different times
  Arms: Group 1
Drug: PF-06473871 — Single dose administered by injection three different times
  Arms: Group 2

SUMMARY:
The study will compare how well PF-06473871 works versus placebo in reducing skin scarring after scar revision surgery of existing breast scars. The study will also evaluate the safety of PF-06473871 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have hypertrophic (raised) breast scars from previous surgery
* Subjects must be healthy

Exclusion Criteria:

* Currently pregnant or pregnant during the 6 months, prior to inclusion in the study or breast-feeding.
* Presence of history of breast cancer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (36):
  - University of California Irvine - Dermatology Research, Irvine, California
  - Plastic Surgery and Laser Institute of San Diego, La Jolla, California
  - Scripps Memorial-Ximed Medical Center, La Jolla, California
  - Advanced Cosmetic Surgery Clinic of Walnut Creek, Walnut Creek, California
  - Anthony DeMeo, MD, Walnut Creek, California
  - Charles Hanson MD, Walnut Creek, California
  - PIH Health Plastic Surgery and Aesthetic Medicine, Whittier, California
  - PIH health, Whittier, California
  - Sanctuary Mediacal Center, Boca Raton, Florida
  - Stephan Baker, MD PA, Coral Gables, Florida
  - Altus Research, Lake Worth, Florida
  - Bayside Ambulatory Center, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Atlanta APC Plastic Surgery, Atlanta, Georgia
  - Kavali Plastic Surgery and Skin Renewal Center, Atlanta, Georgia
  - Perimeter Outpatient Surgery Center, Atlanta, Georgia
  - Advanced Medical Resarch ,Inc, Atlanta, Georgia
  - Atlanta APC Plastic Surgery, Conyers, Georgia
  - Spivey Station Surgery Center, Jonesboro, Georgia
  - Northwestern University Diagnostic Testing Center, Chicago, Illinois
  - Northwestern University,Division of Plastic Surgery, Chicago, Illinois
  - Body Aesthetic Research Center, St Louis, Missouri
  - Mercy Clinic Heart and Vascular, St Louis, Missouri
  - Long Island Plastic Surgical Group, P.C, Garden City, New York
  - Long Island Plastic Surgical Group, P.C., Manhasset, New York
  - Laser Skin Surgery Center of NY, New York, New York
  - The Hunstad Kortesis Center for Cosmetic Surgery, Huntersville, North Carolina
  - Connall Consmetic Surgery, Tualatin, Oregon
  - Meridian Center for Surgical Excellence, LLC, Tualatin, Oregon
  - Timothy P. Connall, MD PC, Tualatin, Oregon
  - Office of Paul M. Glat ,MD, Bala-Cynwyd, Pennsylvania
  - Black Hill Surgical Hospital, Rapid City, South Dakota
  - Health Concepts, Rapid City, South Dakota
  - Fort Bend Imaging, Sugar Land, Texas
  - Luxe Plastic Surgery, Sugar Land, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Noahklinik,Klinik Plastische, Rekonstruktive und Asthetische Chirurgie, Handchirurgie am Roten Kreuz, Kassel, Hesse, Germany
- Magyar Honvedseg-Egeszsegugyi Kozpont, Budapest, Budapest, Hungary
- Spain (2):
  - Hospital Santa Creu I Sant Pau, Barcelona, Barcelona
  - Clinica La Luz, Madrid, Madrid

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5301001&StudyName=Safety%20and%20Efficacy%20Study%20of%20PF-06473871%20to%20Reduce%20Hypertrophic%20Scars%20from%20Recurring%20Post-Revision%20Surgery

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 103 participants were randomized into the study. Of these, 100 participants received at least 1 dose of study drug and were included in the modified intent to treat (mITT) and safety population.
Groups:
- PF-06473871/Placebo (4* 5 mg/cm): Participants with bilateral hypertrophic scars received 4 intradermal injections of PF-06473871 at a dose of 5 milligram per linear centimeter (mg/cm) (2.5 mg on each side of the revised scar) on one breast at Week 2, 5, 8 and 11; and 4 intradermal injections of placebo matched to PF-06473871 at Week 2, 5, 8 and 11 on another breast.
- PF-06473871/Placebo (3* 5 mg/cm): Participants with bilateral hypertrophic scars received 3 intradermal injections of PF-06473871 at a dose of 5 milligrams per linear centimeter (mg/cm) (2.5 mg on each side of the revised scar) on one breast at Week 2, 5 and 8; and 3 intradermal injections of placebo matched to PF-06473871 at Week 2, 5 and 8 on another breast.
Period: Overall Study
Arm/Group | PF-06473871/Placebo (4* 5 mg/cm) | PF-06473871/Placebo (3* 5 mg/cm)
Started | 45 | 55
Completed | 40 | 52
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Un-specified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent To Treat (mITT) population included all participants who were randomized and received at least 1 dose of investigational product.
Groups:
- PF-06473871/Placebo (4* 5 mg/cm): Participants with bilateral hypertrophic scars received 4 intradermal injections of PF-06473871 at a dose of 5 mg/cm ( 2.5 mg on each side of the revised scar) on one breast at Week 2, 5, 8 and 11; and 4 intradermal injections of placebo matched to PF-06473871 at Week 2, 5, 8 and 11 on another breast.
- PF-06473871/Placebo (3* 5 mg/cm): Participants with bilateral hypertrophic scars received 3 intradermal injections of PF-06473871 at a dose of 5 mg/cm (2.5 mg on each side of the revised scar) on one breast at Week 2, 5 and 8; and 3 intradermal injections of placebo matched to PF-06473871 at Week 2, 5 and 8 on another breast.
- Total: Total of all reporting groups
Arm/Group | PF-06473871/Placebo (4* 5 mg/cm) | PF-06473871/Placebo (3* 5 mg/cm) | Total
Number analyzed (Participants) | 45 | 55 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (8.55) | 37.6 (9.64) | 37.9 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 53 | 97
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 39 | 66
  White | 13 | 16 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Pre-Surgery Physician Overall Opinion POSAS Score [Mean (Standard Deviation); unit: units on scale] — Physician global assessment was performed using the overall opinion question of the POSAS scale. Physicians were asked to rate the severity of the participant's scar compared to normal skin. The overall opinion scale score ranged from 1 (normal skin) to 10 (worst imaginable scar).
  units on scale | 6.62 (1.545) | 6.88 (1.277) | 6.76 (1.404)
Pre-Surgery Subject Global Assessment Score [Mean (Standard Deviation); unit: units on scale] — Patient global assessment was performed using the overall opinion question of the POSAS scale. Participants were asked to rate the severity of their scar compared to normal skin. The overall opinion scale score ranged from 1 (normal skin) to 10 (very different from normal skin).
  units on scale | 9.00 (1.219) | 8.49 (1.617) | 8.72 (1.465)
Pre-Surgery Physician Photoguide Score [Mean (Standard Deviation); unit: units on scale] — Physician rated severity of each scar using a photonumeric guide on a scale ranging from 1 to 5 (where 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe).
  units on scale | 3.97 (0.682) | 3.98 (0.725) | 3.98 (0.702)
Pre-Surgery Participant Photoguide Score [Mean (Standard Deviation); unit: units on scale] — Participants rated severity of each scar using a photonumeric guide on a scale ranging from 1 to 5 (where 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe).
  units on scale | 4.24 (0.648) | 4.28 (0.637) | 4.26 (0.639)

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Assessment Using Physician Overall Opinion Question of Patient and Observer Scar Assessment Scale (POSAS)
Description: Physician global assessment was performed using the overall opinion question of the POSAS scale. Physicians were asked to rate the severity of the participant's scar compared to normal skin. The overall opinion scale score ranged from 1 (normal skin) to 10 (worst imaginable scar). Within participant treatment difference was assessed between the treatment regimens each participant received.
Time Frame: Week 24
Population: Modified Intent To Treat (mITT) population included all participants who were randomized and received at least 1 dose of investigational product. Here, N (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Groups:
- Group 1: PF-06473871: 4* 5 mg/cm: Participants with bilateral hypertrophic scars received 4 intradermal injections of PF-06473871 at a dose of 5 mg/cm ( 2.5 mg on each side of the revised scar) on one breast at Week 2, 5, 8, and 11.
- Group 1: Placebo 4* 5 mg/cm: Participants who received 4 intradermal injections of PF-06473871 on one breast and 4 intradermal injections of placebo matched to PF-06473871 at Week 2, 5, 8, and 11 on another breast.
- Group 2: PF¬06473871: 3* 5 mg/cm: Participants with bilateral hypertrophic scars received 3 intradermal injections of PF-06473871 at a dose of 5 mg/cm (2.5 mg on each side of the revised scar) on one breast at Week 2, 5, and 8.
- Group 2: Placebo 3* 5 mg/cm: Participants who received 3 intradermal injections of PF-06473871 on one breast, and 3 intradermal injections of placebo matched to PF-06473871 at Week 2, 5, and 8 on another breast.
Arm/Group | Group 1: PF-06473871: 4* 5 mg/cm | Group 1: Placebo 4* 5 mg/cm | Group 2: PF¬06473871: 3* 5 mg/cm | Group 2: Placebo 3* 5 mg/cm
Number analyzed (Participants) | 43 | 43 | 53 | 53
units on scale | 4.00 (0.30) | 4.68 (0.27) | 4.61 (0.29) | 4.86 (0.28)
Statistical Analysis 1: Comparison: Group 1: PF-06473871: 4* 5 mg/cm vs Group 1: Placebo 4* 5 mg/cm; A total sample size of 100 (accounting for approximately 10% drop rate) that is approximately 50 per group at one sided 0.05 level with delta of 1.5 points with standard deviation of 2 provided at least 80% power to detect a difference from placebo using a paired test. Statistical significance was tested at the two-sided significance level of 0.1, without adjusting for multiplicity; Test type: Superiority or Other; p = 0.0219, Repeated measures model; Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Least Square mean difference = 0.68, 90% CI 2-sided [0.19 to 1.16], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Group 2: PF¬06473871: 3* 5 mg/cm vs Group 2: Placebo 3* 5 mg/cm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4038, Repeated measures model; Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Least Square mean difference = 0.24, 90% CI 2-sided [-0.24 to 0.72], Standard Error of Mean 0.29

2. Secondary Outcome: Physician Scar Assessment Using Complete Patient and Observer Scar Assessment Scale (POSAS)
Description: Physician scar assessment was performed using 10-point POSAS scale. Physician rated each of the items (vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion) for a scar on a score of 1 (normal skin) to 10 (worst scar imaginable). Within participant treatment difference was assessed between the treatment regimens each participant received. Data for overall opinion scale score at Week 24 was not presented in this outcome measure because the data was reported separately under primary outcome measure 1.
Time Frame: Week 8, 11, 18, 24
Population: mITT population included all participants who were randomized and received at least 1 dose of investigational product. Here,"n""= participants who were evaluable at given time point for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Groups:
- Group 1: PF-06473871: (4* 5 mg/cm): Participants with bilateral hypertrophic scars received 4 intradermal injections of PF-06473871 at a dose of 5 mg/cm ( 2.5 mg on each side of the revised scar) on one breast at Week 2, 5, 8, and 11.
- Group 2: PF-06473871: (3* 5 mg/cm): Participants with bilateral hypertrophic scars received 3 intradermal injections of PF-06473871 at a dose of 5 mg/cm (2.5 mg on each side of the revised scar) on one breast at Week 2, 5, and 8.
- Group 2: Placebo 3* 5 mg/cm: Participants who received 3 intradermal injections of PF-06473871 on one breast, also received 3 intradermal injections of placebo matched to PF-06473871 at Week 2, 5, and 8 on another breast.
Arm/Group | Group 1: PF-06473871: (4* 5 mg/cm) | Group 1: Placebo 4* 5 mg/cm | Group 2: PF-06473871: (3* 5 mg/cm) | Group 2: Placebo 3* 5 mg/cm
Number analyzed (Participants) | 45 | 45 | 55 | 55
units on scale
  Vascularity: Week 8 (n=43,43,51,51) | 3.63 (0.24) | 3.51 (0.25) | 3.95 (0.24) | 3.79 (0.24)
  Vascularity: Week 11 (n=43,43,52,52) | 3.64 (0.25) | 3.83 (0.26) | 3.76 (0.26) | 3.83 (0.25)
  Vascularity: Week 18 (n=40,40,52,52) | 3.31 (0.27) | 3.73 (0.28) | 3.49 (0.27) | 3.84 (0.26)
  Vascularity: Week 24 (n=43,43,53,53) | 3.08 (0.27) | 3.40 (0.28) | 3.34 (0.27) | 3.55 (0.27)
  Pigmentation: Week 8 (n=43,43,51,51) | 3.42 (0.23) | 3.53 (0.23) | 3.49 (0.20) | 3.43 (0.19)
  Pigmentation: Week 11 (n=43,43,52,52) | 3.84 (0.27) | 3.73 (0.27) | 3.80 (0.23) | 3.53 (0.22)
  Pigmentation: Week 18 (n=40,40,52,52) | 3.85 (0.29) | 3.88 (0.29) | 3.73 (0.24) | 3.75 (0.23)
  Pigmentation: Week 24 (n=43,43,53,53) | 3.84 (0.29) | 3.99 (0.29) | 4.16 (0.25) | 4.12 (0.24)
  Thickness: Week 8 (n=43,43,51,51) | 3.38 (0.23) | 3.56 (0.24) | 3.59 (0.22) | 3.56 (0.22)
  Thickness: Week 11(n=43,43,52,52) | 3.58 (0.26) | 3.98 (0.26) | 4.01 (0.25) | 3.82 (0.24)
  Thickness: Week 18 (n=40,40,52,52) | 3.67 (0.32) | 4.61 (0.32) | 4.18 (0.30) | 4.39 (0.29)
  Thickness: Week 24 (n=43,43,53,53) | 3.90 (0.32) | 4.58 (0.33) | 4.63 (0.31) | 4.77 (0.30)
  Relief: Week 8 (n=43,43,51,51) | 3.19 (0.23) | 3.58 (0.24) | 3.48 (0.24) | 3.37 (0.22)
  Relief: Week 11(n=43,43,52,52) | 3.63 (0.26) | 3.85 (0.27) | 3.89 (0.27) | 3.70 (0.25)
  Relief: Week 18 (n=40,40,52,52) | 3.75 (0.31) | 4.48 (0.32) | 3.99 (0.31) | 4.08 (0.28)
  Relief: Week 24 (n=43,43,53,53) | 3.87 (0.30) | 4.39 (0.31) | 4.38 (0.29) | 4.53 (0.27)
  Pliability: Week 8 (n=43,43,51,51) | 3.55 (0.25) | 3.84 (0.24) | 3.57 (0.22) | 3.55 (0.21)
  Pliability: Week 11(n=43,43,52,52) | 3.71 (0.28) | 4.02 (0.27) | 4.01 (0.25) | 3.65 (0.24)
  Pliability: Week 18 (n=40,40,52,52) | 3.46 (0.31) | 4.19 (0.30) | 3.86 (0.27) | 3.84 (0.26)
  Pliability: Week 24 (n=43,43,53,53) | 3.73 (0.34) | 4.27 (0.32) | 4.05 (0.30) | 4.54 (0.29)
  Surface Area: Week 8 (n=43,43,51,51) | 3.42 (0.25) | 3.59 (0.23) | 3.48 (0.22) | 3.55 (0.21)
  Surface Area: Week 11 (n=43,43,52,52) | 3.55 (0.27) | 4.06 (0.25) | 3.91 (0.23) | 3.76 (0.22)
  Surface Area: Week 18 (n=40,40,52,52) | 3.97 (0.31) | 4.61 (0.29) | 4.33 (0.26) | 4.32 (0.25)
  Surface Area: Week 24 (n=43,43,53,53) | 4.05 (0.33) | 4.73 (0.30) | 4.55 (0.28) | 4.78 (0.27)
  Overall Opinion: Week 8 (n=43,43,51,51) | 3.50 (0.22) | 3.74 (0.20) | 3.66 (0.22) | 3.75 (0.21)
  Overall Opinion: Week 11 (n=43,43,52,52) | 3.82 (0.25) | 4.05 (0.24) | 4.13 (0.25) | 3.91 (0.24)
  Overall Opinion: Week 18 (n=40,40,52,52) | 3.86 (0.29) | 4.68 (0.27) | 4.35 (0.28) | 4.47 (0.27)
Statistical Analysis 1: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Vascularity: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.12, 90% CI 2-sided [-0.43 to 0.20], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Vascularity: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.16, 90% CI 2-sided [-0.43 to 0.11], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Vascularity: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.19, 90% CI 2-sided [-0.15 to 0.52], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Vascularity: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.07, 90% CI 2-sided [-0.22 to 0.36], Standard Error of Mean 0.17
Statistical Analysis 5: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Vascularity: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.42, 90% CI 2-sided [0.07 to 0.77], Standard Error of Mean 0.21
Statistical Analysis 6: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Vascularity: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.35, 90% CI 2-sided [0.05 to 0.65], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Vascularity: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.33, 90% CI 2-sided [-0.03 to 0.68], Standard Error of Mean 0.21
Statistical Analysis 8: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Vascularity: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.22, 90% CI 2-sided [-0.09 to 0.52], Standard Error of Mean 0.18
Statistical Analysis 9: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Pigmentation: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.12, 90% CI 2-sided [-0.18 to 0.42], Standard Error of Mean 0.18
Statistical Analysis 10: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Pigmentation: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.07, 90% CI 2-sided [-0.35 to 0.22], Standard Error of Mean 0.17
Statistical Analysis 11: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Pigmentation: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.11, 90% CI 2-sided [-0.47 to 0.24], Standard Error of Mean 0.21
Statistical Analysis 12: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Pigmentation: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.27, 90% CI 2-sided [-0.60 to 0.06], Standard Error of Mean 0.20
Statistical Analysis 13: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Pigmentation: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.03, 90% CI 2-sided [-0.35 to 0.41], Standard Error of Mean 0.23
Statistical Analysis 14: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Pigmentation: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.02, 90% CI 2-sided [-0.33 to 0.37], Standard Error of Mean 0.21
Statistical Analysis 15: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Pigmentation: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.14, 90% CI 2-sided [-0.24 to 0.53], Standard Error of Mean 0.23
Statistical Analysis 16: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Pigmentation: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.03, 90% CI 2-sided [-0.39 to 0.32], Standard Error of Mean 0.21
Statistical Analysis 17: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Thickness: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.18, 90% CI 2-sided [-0.22 to 0.58], Standard Error of Mean 0.24
Statistical Analysis 18: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Thickness: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.03, 90% CI 2-sided [-0.42 to 0.35], Standard Error of Mean 0.23
Statistical Analysis 19: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Thickness: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.40, 90% CI 2-sided [-0.05 to 0.84], Standard Error of Mean 0.27
Statistical Analysis 20: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Thickness: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.19, 90% CI 2-sided [-0.62 to 0.23], Standard Error of Mean 0.25
Statistical Analysis 21: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Thickness: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.94, 90% CI 2-sided [0.40 to 1.49], Standard Error of Mean 0.33
Statistical Analysis 22: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Thickness: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.21, 90% CI 2-sided [-0.30 to 0.72], Standard Error of Mean 0.31
Statistical Analysis 23: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Thickness: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.68, 90% CI 2-sided [0.13 to 1.24], Standard Error of Mean 0.34
Statistical Analysis 24: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Thickness: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.14, 90% CI 2-sided [-0.38 to 0.67], Standard Error of Mean 0.32
Statistical Analysis 25: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Relief: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.39, 90% CI 2-sided [-0.01 to 0.78], Standard Error of Mean 0.24
Statistical Analysis 26: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Relief: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.11, 90% CI 2-sided [-0.50 to 0.28], Standard Error of Mean 0.23
Statistical Analysis 27: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Relief: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.22, 90% CI 2-sided [-0.23 to 0.67], Standard Error of Mean 0.27
Statistical Analysis 28: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Relief: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.19, 90% CI 2-sided [-0.63 to 0.24], Standard Error of Mean 0.26
Statistical Analysis 29: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Relief: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.74, 90% CI 2-sided [0.21 to 1.26], Standard Error of Mean 0.31
Statistical Analysis 30: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Relief: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.09, 90% CI 2-sided [-0.41 to 0.59], Standard Error of Mean 0.30
Statistical Analysis 31: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Relief: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.52, 90% CI 2-sided [0.02 to 1.02], Standard Error of Mean 0.30
Statistical Analysis 32: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Relief: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.15, 90% CI 2-sided [-0.33 to 0.63], Standard Error of Mean 0.29
Statistical Analysis 33: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Pliability: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.29, 90% CI 2-sided [-0.09 to 0.67], Standard Error of Mean 0.23
Statistical Analysis 34: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Pliability: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.03, 90% CI 2-sided [-0.39 to 0.34], Standard Error of Mean 0.22
Statistical Analysis 35: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Pliability: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.31, 90% CI 2-sided [-0.12 to 0.74], Standard Error of Mean 0.26
Statistical Analysis 36: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Pliability: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.35, 90% CI 2-sided [-0.76 to 0.05], Standard Error of Mean 0.25
Statistical Analysis 37: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Pliability: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.73, 90% CI 2-sided [0.25 to 1.20], Standard Error of Mean 0.29
Statistical Analysis 38: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Pliability: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.02, 90% CI 2-sided [-0.46 to 0.42], Standard Error of Mean 0.27
Statistical Analysis 39: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Pliability: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.53, 90% CI 2-sided [0.01 to 1.05], Standard Error of Mean 0.31
Statistical Analysis 40: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Pliability: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.49, 90% CI 2-sided [0.00 to 0.98], Standard Error of Mean 0.30
Statistical Analysis 41: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Surface Area: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.17, 90% CI 2-sided [-0.29 to 0.62], Standard Error of Mean 0.27
Statistical Analysis 42: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Surface Area: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.08, 90% CI 2-sided [-0.28 to 0.43], Standard Error of Mean 0.21
Statistical Analysis 43: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Surface Area: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.51, 90% CI 2-sided [0.02 to 1.00], Standard Error of Mean 0.30
Statistical Analysis 44: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Surface Area: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.15, 90% CI 2-sided [-0.53 to 0.23], Standard Error of Mean 0.23
Statistical Analysis 45: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Surface Area: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.64, 90% CI 2-sided [0.08 to 1.20], Standard Error of Mean 0.34
Statistical Analysis 46: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Surface Area : Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.01, 90% CI 2-sided [-0.44 to 0.42], Standard Error of Mean 0.26
Statistical Analysis 47: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Surface Area: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.69, 90% CI 2-sided [0.09 to 1.28], Standard Error of Mean 0.36
Statistical Analysis 48: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Surface Area: week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.23, 90% CI 2-sided [-0.23 to 0.69], Standard Error of Mean 0.28
Statistical Analysis 49: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Overall Opinion: Week 8 A total sample size of 100 (accounting for approximately 10% drop rate) that is approximately 50 per group at one sided 0.05 level with delta of 1.5 points with standard deviation of 2 provided at least 80% power to detect a difference from placebo using a paired test. Statistical significance was tested at the two-sided significance level of 0.1, without adjusting for multiplicity; Test type: Superiority or Other; p = 0.2778, Repeated measures model; Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Least Square mean difference = 0.24, 90% CI 2-sided [-0.12 to 0.60], Standard Error of Mean 0.22
Statistical Analysis 50: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Overall Opinion: Weekl 8 A total sample size of 100 (accounting for approximately 10% drop rate) that is approximately 50 per group at one sided 0.05 level with delta of 1.5 points with standard deviation of 2 provided at least 80% power to detect a difference from placebo using a paired test. Statistical significance was tested at the two-sided significance level of 0.1, without adjusting for multiplicity; Test type: Superiority or Other; p = 0.6888, Repeated measures model; Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Least Square mean difference = 0.09, 90% CI 2-sided [-0.28 to 0.45], Standard Error of Mean 0.22
Statistical Analysis 51: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Overall Opinion: Weekl 11 A total sample size of 100 (accounting for approximately 10% drop rate) that is approximately 50 per group at one sided 0.05 level with delta of 1.5 points with standard deviation of 2 provided at least 80% power to detect a difference from placebo using a paired test. Statistical significance was tested at the two-sided significance level of 0.1, without adjusting for multiplicity; Test type: Superiority or Other; p = 0.3515, Repeated measures model; Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Least Square mean difference = 0.23, 90% CI 2-sided [-0.18 to 0.65], Standard Error of Mean 0.25
Statistical Analysis 52: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; [analysis description as in outcome 2, analysis 51]; Test type: Superiority or Other; p = 0.3788, Repeated measures model; Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Least Square mean difference = -0.22, 90% CI 2-sided [-0.64 to 0.19], Standard Error of Mean 0.25
Statistical Analysis 53: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Overall Opinion: Weekl 18 A total sample size of 100 (accounting for approximately 10% drop rate) that is approximately 50 per group at one sided 0.05 level with delta of 1.5 points with standard deviation of 2 provided at least 80% power to detect a difference from placebo using a paired test. Statistical significance was tested at the two-sided significance level of 0.1, without adjusting for multiplicity; Test type: Superiority or Other; p = 0.0044, Repeated measures model; Least Square mean difference = 0.82, 90% CI 2-sided [0.35 to 1.29], Standard Error of Mean 0.28
Statistical Analysis 54: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; [analysis description as in outcome 2, analysis 53]; Test type: Superiority or Other; p = 0.6848, Repeated measures model; Least Square mean difference = 0.11, 90% CI 2-sided [-0.35 to 0.58], Standard Error of Mean 0.28

3. Secondary Outcome: Patient Global Assessment Using Overall Opinion of Patient and Observer Scar Assessment Scale (POSAS)
Description: Patient global assessment was performed using the overall opinion question of the POSAS scale. Participants were asked to rate the severity of their scar compared to normal skin. The overall opinion scale score ranged from 1 (normal skin) to 10 (very different from normal skin). Within participant treatment difference was assessed between the treatment regimens each participant received
Time Frame: Week 8, 11, 18, 24
Population: mITT population included all participants who were randomized and received at least 1 dose of investigational product. Here, "n""= participants who were evaluable at given time point for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Groups:
- Group 1: Placebo 4* 5 mg/cm: Participants who received 4 intradermal injections of PF-06473871 on one breast, and 4 intradermal injections of placebo matched to PF-06473871 at Week 2, 5, 8, and 11 on another breast.
Arm/Group | Group 1: PF-06473871: (4* 5 mg/cm) | Group 1: Placebo 4* 5 mg/cm | Group 2: PF-06473871: (3* 5 mg/cm) | Group 2: Placebo 3* 5 mg/cm
Number analyzed (Participants) | 45 | 45 | 55 | 55
units on scale
  Week 8: (n=43,43,51,51) | 5.38 (0.33) | 5.48 (0.31) | 5.09 (0.32) | 5.20 (0.29)
  Week 11: (n=43,43,52,52) | 5.58 (0.33) | 5.59 (0.32) | 4.52 (0.32) | 4.73 (0.30)
  Week 18: (n=40,40,52,52) | 5.34 (0.38) | 5.78 (0.36) | 5.18 (0.36) | 5.18 (0.33)
  Week 24: (n=43,43,53,53) | 5.65 (0.39) | 5.94 (0.37) | 5.33 (0.38) | 5.15 (0.35)
Statistical Analysis 1: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; p = 0.7552, Repeated measures model; Least Square mean difference = 0.10, 90% CI 2-sided [-0.44 to 0.64], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; p = 0.6605, Repeated measures model; LS mean difference = 0.11, 90% CI 2-sided [-0.30 to 0.52], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; p = 0.9842, Repeated measures model; Least Square mean difference = 0.01, 90% CI 2-sided [-0.55 to 0.56], Standard Error of Mean 0.33
Statistical Analysis 4: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; p = 0.4010, Repeated measures model; Least Square mean difference = 0.21, 90% CI 2-sided [-0.21 to 0.63], Standard Error of Mean 0.25
Statistical Analysis 5: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; p = 0.2491, Repeated measures model; Least Square mean difference = 0.44, 90% CI 2-sided [-0.19 to 1.07], Standard Error of Mean 0.38
Statistical Analysis 6: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; p = 0.9980, Repeated measures model; Least Square mean difference = 0.00, 90% CI 2-sided [-0.47 to 0.47], Standard Error of Mean 0.29
Statistical Analysis 7: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; p = 0.4730, Repeated measures model; Least Square mean difference = 0.28, 90% CI 2-sided [-0.37 to 0.93], Standard Error of Mean 0.39
Statistical Analysis 8: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; p = 0.5413, Repeated measures model; Least Square mean difference = -0.18, 90% CI 2-sided [-0.67 to 0.31], Standard Error of Mean 0.30

4. Secondary Outcome: Patient-Reported Scar Evaluation Questionnaire (PR-SEQ) Symptoms and Appearance Domains Score
Description: PR-SEQ questionnaire consisted of 30 different attributes of scars that included following four dimensions: appearance (5 attributes), symptoms (3 attributes), bothersomeness (8 attributes), and impacts on the quality of life (physical and emotional wellbeing [14 attributes]). Each question had 5 possible responses: not at all (0), slightly (1), moderately (2), very (3), and extremely (4). Participants completed an abbreviated version which included only the Symptoms and Appearance dimensions to evaluate treatment outcomes. Each of the item scores were transformed into a 0 to 100 scale. Each dimension score was calculated from averaging the transformed scores (0-100 scaled) for specified items. Each domain score ranged from 0 to 100, with higher scores indicating higher severity. Within participant treatment difference was assessed between the treatment regimens each participant received.
Time Frame: Week 8, 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Group 1: PF-06473871: (4* 5 mg/cm) | Group 1: Placebo 4* 5 mg/cm | Group 2: PF-06473871: (3* 5 mg/cm) | Group 2: Placebo 3* 5 mg/cm
Number analyzed (Participants) | 45 | 45 | 55 | 55
units on scale
  Appearance: Week 8: (n=43,43,53,53) | 34.95 (2.38) | 36.27 (2.27) | 34.50 (2.20) | 34.14 (2.20)
  Appearance: Week 24: (n=43,43,54,54) | 43.55 (3.32) | 47.37 (3.16) | 42.41 (3.04) | 42.56 (3.04)
  Symptoms: Week 8: (n=43,43,53,53) | 17.89 (2.62) | 17.19 (2.34) | 18.46 (2.71) | 16.92 (2.47)
  Symptoms: Week 24: (n=43,43,54,54) | 13.74 (2.75) | 15.49 (2.45) | 18.22 (2.81) | 17.09 (2.57)
Statistical Analysis 1: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Appearance: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 1.32, 90% CI 2-sided [-3.28 to 5.92], Standard Error of Mean 2.76
Statistical Analysis 2: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Appearance: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; LS mean difference = -0.36, 90% CI 2-sided [-3.63 to 2.91], Standard Error of Mean 1.97
Statistical Analysis 3: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Appearance: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 3.82, 90% CI 2-sided [-2.60 to 10.24], Standard Error of Mean 3.85
Statistical Analysis 4: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Appearance: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.16, 90% CI 2-sided [-4.37 to 4.68], Standard Error of Mean 2.72
Statistical Analysis 5: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Symptoms: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.70, 90% CI 2-sided [-4.34 to 2.95], Standard Error of Mean 2.19
Statistical Analysis 6: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Symptoms: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -1.54, 90% CI 2-sided [-4.53 to 1.45], Standard Error of Mean 1.80
Statistical Analysis 7: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Symptoms: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 1.75, 90% CI 2-sided [-2.07 to 5.58], Standard Error of Mean 2.30
Statistical Analysis 8: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Symptoms: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -1.13, 90% CI 2-sided [-4.24 to 1.99], Standard Error of Mean 1.87

5. Secondary Outcome: Physician and Participant Photoguide Scar Assessment Scale Score
Description: Physician and participants rated severity of each scar using a photonumeric guide on a scale ranging from 1 to 5 (where 1 = minimal, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe). Within participant treatment difference was assessed between the treatment regimens each participant received.
Time Frame: Week 8, 11, 18, 24
Population: mITT population included all participants who were randomized and received at least 1 dose of investigational product. Here, "n"= participants who were evaluable at given time point for each arm, respectively.
Measure: Least Squares Mean (Standard Error); unit: units on scale
Arm/Group | Group 1: PF-06473871: (4* 5 mg/cm) | Group 1: Placebo 4* 5 mg/cm | Group 2: PF-06473871: (3* 5 mg/cm) | Group 2: Placebo 3* 5 mg/cm
Number analyzed (Participants) | 45 | 45 | 55 | 55
units on scale
  Physician: Week 8 (n=43,43,52,52) | 2.35 (0.15) | 2.45 (0.14) | 2.24 (0.16) | 2.28 (0.14)
  Physician: Week 11 (n=43,43,53,53) | 2.42 (0.15) | 2.71 (0.14) | 2.58 (0.16) | 2.48 (0.14)
  Physician: Week 18 (n=40,40,53,53) | 2.48 (0.15) | 3.05 (0.14) | 2.70 (0.16) | 2.74 (0.14)
  Physician: Week 24 (n=43,43,54,54) | 2.60 (0.15) | 3.03 (0.14) | 3.00 (0.16) | 3.07 (0.14)
  Participant: Week 8 (n=43,43,52,52) | 2.41 (0.16) | 2.51 (0.16) | 2.28 (0.15) | 2.25 (0.14)
  Participant: Week 11 (n=43,43,53,53) | 2.65 (0.16) | 2.66 (0.16) | 2.48 (0.15) | 2.56 (0.14)
  Participant: Week 18 (n=39,39,53,53) | 2.38 (0.16) | 2.80 (0.17) | 2.80 (0.15) | 2.79 (0.14)
  Participant: Week 24 (n=43,43,54,54) | 2.75 (0.16) | 2.95 (0.16) | 2.75 (0.15) | 2.89 (0.14)
Statistical Analysis 1: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Physician: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.10, 90% CI 2-sided [-0.15 to 0.35], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Physician: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.03, 90% CI 2-sided [-0.22 to 0.29], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Physician: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.29, 90% CI 2-sided [0.04 to 0.54], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Physician: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.10, 90% CI 2-sided [-0.36 to 0.15], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Physician: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.57, 90% CI 2-sided [0.32 to 0.82], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Physician: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.05, 90% CI 2-sided [-0.21 to 0.30], Standard Error of Mean 0.15
Statistical Analysis 7: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Physician: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.43, 90% CI 2-sided [0.18 to 0.68], Standard Error of Mean 0.15
Statistical Analysis 8: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Physician: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.07, 90% CI 2-sided [-0.18 to 0.32], Standard Deviation 0.15
Statistical Analysis 9: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Participant: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.10, 90% CI 2-sided [-0.20 to 0.39], Standard Error of Mean 0.18
Statistical Analysis 10: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Participant: Week 8: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.02, 90% CI 2-sided [-0.28 to 0.23], Standard Error of Mean 0.15
Statistical Analysis 11: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Participant: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.00, 90% CI 2-sided [-0.29 to 0.30], Standard Error of Mean 0.18
Statistical Analysis 12: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Participant: Week 11: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.07, 90% CI 2-sided [-0.18 to 0.33], Standard Error of Mean 0.15
Statistical Analysis 13: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Participant: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.42, 90% CI 2-sided [0.12 to 0.72], Standard Error of Mean 0.18
Statistical Analysis 14: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Participant: Week 18: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = -0.01, 90% CI 2-sided [-0.27 to 0.24], Standard Error of Mean 0.15
Statistical Analysis 15: Comparison: Group 1: PF-06473871: (4* 5 mg/cm) vs Group 1: Placebo 4* 5 mg/cm; Participant: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.20, 90% CI 2-sided [-0.09 to 0.50], Standard Error of Mean 0.18
Statistical Analysis 16: Comparison: Group 2: PF-06473871: (3* 5 mg/cm) vs Group 2: Placebo 3* 5 mg/cm; Participant: Week 24: Difference is calculated as Placebo minus PF-06473871. A positive difference favors PF-06473871; Test type: Superiority or Other; Least Square mean difference = 0.15, 90% CI 2-sided [-0.11 to 0.40], Standard Error of Mean 0.15

6. Other Pre Specified Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Vital Sign included pulse rate, systolic blood pressure, diastolic blood pressure, and weight.
Time Frame: Baseline up to Week 24
Population: Safety population included all participants who received at least 1 dose of investigational product.
Measure: Number; unit: participants
Groups:
- PF-06473871/Placebo (4* 5 mg/cm): Participants with bilateral hypertrophic scars received 4 intradermal injections of PF-06473871 at a dose of 5 mg/cm, (2.5 mg on each side of the revised scar) on one breast at Week 2, 5, 8 and 11; and 4 intradermal injections of placebo matched to PF-06473871 at Week 2, 5, 8 and 11 on another breast.
Arm/Group | PF-06473871/Placebo (4* 5 mg/cm) | PF-06473871/Placebo (3* 5 mg/cm)
Number analyzed (Participants) | 45 | 55
participants | 0 (0.39) | 0 (0.37)

7. Other Pre Specified Outcome: Number of Participants With Abnormal Physical Examinations
Description: Physical examination included examination of skin, head, eyes, ears, nose, throat (HEENT), respiratory, cardiovascular, abdomen - liver and kidney, musculoskeletal, gastrointestinal, genitourinary, and neurological systems.
Time Frame: Baseline up to Week 24
Population: Safety population included all participants who received at least 1 dose of investigational product.
Measure: Number; unit: participants
Groups:
- PF-06473871/Placebo (4* 5 mg/cm): Participants with bilateral hypertrophic scars received 4 intradermal injections of PF-06473871 at a dose of 5 mg/cm (2.5 mg on each side of the revised scar) on one breast at Week 2, 5, 8 and 11; and 4 intradermal injections of placebo matched to PF-06473871 at Week 2, 5, 8 and 11 on another breast.
Arm/Group | PF-06473871/Placebo (4* 5 mg/cm) | PF-06473871/Placebo (3* 5 mg/cm)
Number analyzed (Participants) | 45 | 55
participants | 0 (0.39) | 0 (0.37)

8. Other Pre Specified Outcome: Number of Participants With Electrocardiogram Findings
Description: Following parameters were assessed: heart rate, PR Interval, QRS Interval, QT Interval, and Fridericia's Correction Formula (QTcF) interval. Electrocardiogram Results were reported as normal, abnormal, not clinically significant (NCS) and abnormal and clinically significant (CS) as determined by investigator.
Time Frame: Baseline, Week 11
Population: Safety population included all participants who received at least 1 dose of investigational product. Here, "n""= participants who were evaluable at given time point for each arm, respectively.
Measure: Number; unit: participants
Arm/Group | PF-06473871/Placebo (4* 5 mg/cm) | PF-06473871/Placebo (3* 5 mg/cm)
Number analyzed (Participants) | 45 | 55
participants
  Baseline: Normal (n=45,55) | 38 (0.39) | 43 (0.37)
  Baseline: Abnormal, NCS (n=45,55) | 7 | 12
  Baseline: Abnormal , CS (n=45,55) | 0 | 0
  Week 11: Normal (n=42,53) | 33 | 43
  Week 11: Abnormal, NCS (n=42,53) | 9 | 10
  Week 11: Abnormal, CS (n=42,53) | 0 | 0

9. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) of Special Interest
Description: Treatment Emergent Adverse Events (AEs) of special interest included injection site erythema, maculopapular rash, pruritus, bronchospasm, dyspnea, cough, fever and diarrhea.
Time Frame: Baseline up to Week 24
Population: Safety population included all participants who received at least 1 dose of investigational product. Here, "N" (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | PF-06473871/Placebo (4* 5 mg/cm) | PF-06473871/Placebo (3* 5 mg/cm)
Number analyzed (Participants) | 45 | 55
participants | 3 (0.39) | 9 (0.37)

10. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Related to Laboratory Abnormalities
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent adverse event are events between first dose of study drug and up to Week 24 that were absent before treatment or that worsened relative to pre-treatment state. TEAEs related to laboratory abnormalities are reported.
Time Frame: Baseline up to Week 24
Population: Safety population included all participants who received at least 1 dose of investigational product.
Measure: Number; unit: participants
Arm/Group | PF-06473871/Placebo (4* 5 mg/cm) | PF-06473871/Placebo (3* 5 mg/cm)
Number analyzed (Participants) | 45 | 55
participants
  Leukopenia | 0 (0.39) | 1 (0.37)
  Hyperbilrubinemia | 0 | 1
  Amylase increased | 1 | 1
  Blood creatine phosphokinase (CPK) increased | 2 | 6
  Blood glucose increased | 0 | 1
  Blood lactate dehydrogenase (LDH) increased | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: There was no overall separate placebo group for safety assessment as each participant received both placebo as well as active drug. AE assessment was done between those who received 3 versus 4 doses of active drug.
Arm/Group | PF-06473871/Placebo (4* 5 mg/cm) | PF-06473871/Placebo (3* 5 mg/cm)
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/55
Other Adverse Events (participants affected / at risk) | 30/45 | 35/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06473871/Placebo (4* 5 mg/cm) (N=45) | PF-06473871/Placebo (3* 5 mg/cm) (N=55)
Injection site erythema (General disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 5 | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 4 | 0
Incision site pruritus (Injury, poisoning and procedural complications) | 1 | 2
Procedural site reaction (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 1 | 0
Incision site blister (Injury, poisoning and procedural complications) | 0 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0
Injection site pain (General disorders) | 10 | 9
Injection site pruritus (General disorders) | 3 | 4
Application site rash (General disorders) | 0 | 1
Injection site rash (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Injection site urticaria (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Viral rhinitis (Infections and infestations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 6
Amylase increased (Investigations) | 1 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 2 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Piriformis syndrome (Nervous system disorders) | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 2
Itching scar (Skin and subcutaneous tissue disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Breast haematoma (Reproductive system and breast disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Treatment noncompliance (Social circumstances) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.